CLINICAL TRIAL: NCT03566381
Title: Pilot Study of a Wearable Sweat Sensor for Hydration Monitoring of Athletes
Brief Title: Sweat Sensors for Athletic Performance
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Instructor, Northwestern University
Other Study IDs: SX01262018
Record Dates: First submitted 2018-05-02; First posted 2018-06-25 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Healthy Adults
Keywords: Wearable sensor, sweat sensor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy adults without a history of medical or surgical problems
  Interventions: Device: Application of a soft patch composed of medical-grade silicone that collects sweat during a subject's natural behaviors.

INTERVENTIONS:
Device: Application of a soft patch composed of medical-grade silicone that collects sweat during a subject's natural behaviors. — This device contains sweat sensors embedded in an elastomer and is applied to the skin with a medical grade adhesive.

SUMMARY:
Pilot study of a soft, flexible wearable sweat sensor

DETAILED DESCRIPTION:
Assessment of safety, and preliminary accuracy of a sweat sensor capable of operating underwater.

ELIGIBILITY:
Inclusion Criteria:

* No history of medical or surgical problems
* Age >18 years old
* Subjects willing and able to comply with requirements of the protocol

Exclusion Criteria:

* Age <18 years old
* Subjects unwilling and able to comply with requirements of the protocol
* History of skin allergy to medical adhesive tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Adhesion of device underwater | 2 hours
  Percentage of devices which remain adhered during >1 hr swim trials

SECONDARY OUTCOMES:
Correlation between local and global sweat loss | 2 hours
  Percentage agreement of local sweat rate with body weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States